CLINICAL TRIAL: NCT07171294
Title: Prospective Observational Study to Assess the Reproducibility of Minimally Invasive Surgery in the Treatment of Grade III Hemorrhoids: Phase 2A of the IDEAL Framework
Brief Title: Reproducibility of Minimally Invasive Surgery for Grade III Hemorrhoids
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Son Llatzer (Other)
Collaborators: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Principal Investigator, Ignacio Fernandez Hurtado, Principal Investigator, Hospital Son Llatzer
Other Study IDs: HEM IDEAL 2A
Record Dates: First submitted 2025-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hemorrhoidectomy; Minimal Invasive Surgery
Keywords: Hemorrhoids grade III-IV; Hemorrhoidectomy; Minimal Invasive Surgery; IDEAL Stage 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Grade III Hemorrhoids: Patients with symptomatic grade III hemorrhoids who consent to surgical interv
  Interventions: Procedure: Minimal invasive hemorrhoidectomy

INTERVENTIONS:
Procedure: Minimal invasive hemorrhoidectomy — We propose applying minimally invasive surgery in open excisional hemorrhoidectomy, the most effective technique for treating advanced hemorrhoidal disease. We believe this approach will reduce postoperative pain and improve recovery while maintaining the excellent outcomes of OEH. Our hypothesis is based on the reduced tissue trauma and increased precision provided by minimally invasive surgery.

SUMMARY:
Hemorrhoids are vascular-elastic structures of the anal canal that contribute to continence. Their enlargement and descent lead to symptoms such as rectal bleeding and the sensation of anal swelling, known as hemorrhoidal syndrome. In advanced cases (Goligher Grade III-IV), surgery is the only effective treatment. Open excisional hemorrhoidectomy (OEH), based on the Milligan-Morgan technique, is the standard procedure. Although effective in the long term, it causes severe postoperative pain. Minimally invasive surgery (MIS) employs enhanced visualization devices to improve surgical precision and reduce tissue damage. While widely used in specialties with small surgical fields, it has not yet been explored in anal surgery. Its advantages include reduced tissue injury and improved healing, although it presents a learning curve and an initially longer surgical time. The IDEAL framework evaluates surgical innovations in five stages: Idea, Development, Exploration, Evaluation, and Long-Term Study. The IDEAL phase 2a is aimed at the optimization and technical definition of surgical innovation with a focus on continuous improvement based on real clinical practice, laying the foundation for broader and more rigorous subsequent studies.

Since no previous studies on the application of MIS in OEH have been found, the investigators propose a study within Stage 2A of the IDEAL model to assess the reproducibility of this technique. The investigators believe its incorporation into open excisional hemorrhoidectomy could result in less postoperative pain and faster patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Grade III hemorrhoids
* BMI below 30
* Indication for OEH surgery
* Signed written informed consent

Exclusion Criteria:

* Acute hemorrhoidal disease (thrombosis)
* Previous hemorrhoid surgery
* Coexistence of anal fissure
* Coexistence of perianal fistula
* Coexistence of rectal or anal prolapse
* Active inflammatory bowel disease
* Active anal or colorectal cancer
* Language barrier or difficulty in oral and/or written comprehension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the Surgery Department of our Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Technical Reproducibility of Surgery | 30 postoperative days
  Since no studies using this approach were found in the literature, the investigators propose a study to assess the reproducibility of implementing this technique following the guidelines of the IDEAL framework. In this study, the investigators propose Stage 2A. The measurement tool will be the systematic documentation of technical modifications.

SECONDARY OUTCOMES:
Adverse events in treated patients | 30 postoperative days
  Collect the adverse effects that occur during the operative period and within the first 30 postoperative days. Filter those attributable to the use of the minimally invasive approach. Analyze the causes and the technical steps that should be performed or omitted to avoid them. As measurement tools, the Clavien-Dindo scale and the Comprehensive Complication Index (CCI) will be used. The CCI is an index that uses the Clavien-Dindo scale and is calculated with a mathematical formula available at www.assessurgery.com
Postoperative pain | The first 14 postoperative days
  Postoperative pain will be evaluated using the Visual Analogue Scale (VAS), a validated tool ranging from 0 (no pain) to 10 (worst imaginable pain). Patients will self-assess their baseline pain and pain following defecation at predefined intervals: postoperative days 4, 7, and 14.
Hemorrhoidal disease symptom score | one postoperative year
  A score that defines the frecuency of pain, pruritus, bleeding, soiling and prolapse. Score 0 to 20. Higher scores mean a worse outcome.
Short Health Scale in hemorrhoidal disease | One year postoperative
  A subjective scale which defines symptom intensity, the patient's worrying and the role in impairment of daily activity. Score 4 to 28. Higher scores mean a worse outcome.
Total number of postoperative analgesics | 14 postoperative days
  The total number of analgesic doses taken by the patient during the first 14 postoperative days will be recorded as a numeric variable

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Son Llatzer, Palma, Spain

IPD SHARING:
Plan to Share IPD: Undecided